CLINICAL TRIAL: NCT03688880
Title: A Randomized, Open-label, Multi-center, Controlled Clinical Study to Compare MAR-CUTIS With Dermabond Advanced in Closure of Surgical Incisions and Lacerations up to 15 Centimeters
Brief Title: A Clinical Study to Compare MAR-CUTIS With Dermabond Advanced
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF7021-04; 1012937 (Other: Syneos Health)
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-07

CONDITIONS: Wounds and Injuries; Lacerations; Surgical Incision
Keywords: Wounds; Injuries; Surgery; Lacerations; Wound healing; Surgical Wounds
MeSH Terms: conditions — Wounds and Injuries; Lacerations; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Dermabond Advanced (Active Comparator): Dermabond Advanced (a topical skin adhesive) was applied on Day 0. Dermabond Advanced was applied in 1 continuous layer onto a dry wound through painting motions; the wound was held for 60 seconds to allow for complete polymerization.
  Interventions: Device: Dermabond Advanced
- MAR-CUTIS (Experimental): MAR-CUTIS (polyurethane-based skin adhesive) was applied on Day 0. MAR-CUTIS was applied in 1 to 2 millimeter (mm) thick layer ensuring that at least 1 cm of the glue is applied over the length of the wound on each side; the wound was held for approximately 30 seconds to allow for initial polymerization.
  Interventions: Device: MAR-CUTIS

INTERVENTIONS:
Device: MAR-CUTIS — MAR-CUTIS was applied in 1 to 2 mm thick layer, ensuring that at least 1 cm of the glue was applied over the length of the wound on each side. The amount of the glue applied was calculated such that one 5-mL syringe covers approximately 8 cm of wound length (giving a total of 10 cm per syringe). For wounds >8 cm, 2 syringes were required.
  Arms: MAR-CUTIS
Device: Dermabond Advanced — Dermabond Advanced was applied in 1 continuous layer onto a dry wound through painting motions, taking care not to apply adhesive between the wound edges.
  Arms: Dermabond Advanced

SUMMARY:
This was a randomized, open-label, multicenter, comparator-controlled clinical study to compare MAR-CUTIS with Dermabond Advanced in closure of surgical incisions and lacerations less than or equal to (<=)15 centimeter (cm). Eligible participants were randomized 2:1 to MAR-CUTIS or Dermabond Advanced.

ELIGIBILITY:
Inclusion Criteria:

For participants with surgical incisions:

1. Participants underwent closure of surgical incision 6 to 15 centimeters (cms) following laparotomy, abdominal hysterectomy, or laparoscopic intervention.

   For participants with lacerations:
2. Participants requiring closure of a laceration on face (avoiding the immediate area around the eye) or extremities. In participants with multiple lacerations, one was selected as the target wound (i.e., greatest length and meets the study entry criteria).

   For all participants:
3. Participant had given written informed consent/assent to participate.
4. Male and female participants at least 2 years of age and body weight 10 kilogram (kg) or greater.
5. Participants willing and capable of following instructions for wound care provided by the investigator and agreeing to return for all treatment control visits specified in this clinical study.

Exclusion Criteria:

For participants with lacerations:

1. Wounds on mucosal surfaces or across mucocutaneous junctions (e.g., oral cavity, lips, eyes).
2. Wounds which might be regularly exposed to body fluids or with dense natural hair (e.g., scalp); wounds on ears.
3. Wounds on palms and feet.
4. Animal or human bites.
5. Lacerations that were heavily contaminated.
6. Punctured or crushed wounds.
7. Participants with lacerations having wound treatment more than 6 hours after the trauma.

   For all participants:
8. Participants requiring suturing with sutures greater than 5 mm thickness.
9. Participants with documented skin disease or skin conditions (e.g., excessive hair at the site of surgery, scar tissue, wound, tattoo, coloration, or pre-existing open sores at the site of surgery that would interfere with the application of Investigational Medical Device or the skin assessment, as judged by the investigator).
10. Participant with any factors that might had an adverse effect on wound healing (e.g., previous history of keloid formation or hypertrophy [as well in the family]), history of immunosuppression, chronic systemic infection, or poor general health.
11. Participants with known blood clotting disorders.
12. Participants receiving steroids, immunosuppressants, chemotherapy, or anticoagulants.
13. Participants having known or suspected allergy or sensitivity to polyurethane, cyanoacrylates, formaldehyde, tapes or adhesives, or benzalkonium chloride.
14. Participant participating in any current clinical study with a non-CE ("Conformitee Europeene") marked device or investigational product.
15. Participant who was pregnant or breastfeeding.
16. Participant with history of a significant dermatologic disease or condition, such as atopic dermatitis, psoriasis, lichen ruber planus, vitiligo or conditions known to alter the skin appearance or physiologic response (e.g., decompensated diabetes mellitus, porphyria) that involves the investigative site.

Removal of Participants From Therapy or Assessments:

Only participants that were withdrawn from the study due to product failure at the time of application were replaced.

Participants might stop the study for any of the following reasons:

1. Participant request.
2. Use of non-permitted concurrent therapy.
3. Lost to follow-up (considered lost to follow-up only before Day 10).
4. Occurrence of adverse events not compatible with the continuation of participant participation in the study, in the investigator's opinion, or unacceptable to the participant to continue.

   * Investigator request.
   * Inter-current illness.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH
Locations (19):
- France (2):
  - 004 - CHU Amiens-Picardie, Amiens
  - 005 - Hôpital Privé Paul d'Egine, Champigny-sur-Marne
- Germany (3):
  - 010 - Charité Berlin, Berlin
  - 006 - Universitätsklinikum Heidelberg, Heidelberg
  - 009 - Klinikum Magdeburg, Magdeburg
- Spain (3):
  - 001 - Hospital Universitari Vall d'Hebron, Barcelona
  - 022 - Hospital General Universitario Gregorio Maranon, Madrid
  - 003 - University Hospital Virgen del Rocío, Seville
- United Kingdom (11):
  - 019 - Barnsley Hospital, Barnsley
  - 017 - Birmingham Children's Hospital, Birmingham
  - 018 - Bristol Royal Hospital for Children, Bristol
  - 021 - University Hospital of Wales, Cardiff
  - 013 - The Princess Alexandra Hospital, Harlow
  - 011 - Leeds Teaching Hospitals, Leeds
  - 016 - St George's Hospital, London
  - 014 - Queen Elizabeth the Queen Mother Hospital, Margate
  - 020 - Royal Gwent Hospital, Newport
  - 012 - Peterborough City Hospital, Peterborough
  - 015 - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 sites in 4 countries from 30 October 2018 to 04 September 2019. A total of 107 participants were enrolled of which 18 participants were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: A Total of 89 participants were randomized and treated in the study. Assignment to arms was done in 2:1 ratio (MAR-CUTIS:Dermabond Advanced). Randomization was stratified by wound type (lacerations and incisions), skin type and age groups.
Period: Overall Study
Arm/Group | Dermabond Advanced | MAR-CUTIS
Started | 29 | 60
Completed | 15 | 29
Not Completed | 14 | 31
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Use of non-permitted concurrent therapy | 0 | 2
Not completed — Lost to Follow-up | 4 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Device deficiencies | 0 | 2
Not completed — Other | 10 | 16

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety analysis set which included all participants where the application of MAR-CUTIS or Dermabond Advanced had started. Participants were analyzed under the actual treatment received.
Groups:
- MAR-CUTIS: MAR-CUTIS (polyurethane-based skin adhesive) was applied on Day 0. MAR-CUTIS was applied in 1 to 2 mm thick layer ensuring that at least 1 cm of the glue is applied over the length of the wound on each side; the wound was held for approximately 30 seconds to allow for initial polymerization.
- Total: Total of all reporting groups
Arm/Group | Dermabond Advanced | MAR-CUTIS | Total
Number analyzed (Participants) | 29 | 60 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (26.7) | 49.9 (24.9) | 48.3 (25.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 25 | 34
  Male | 20 | 35 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 27 | 55 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Dehiscence of Target Wound at Day 10
Description: Wound dehiscence involved the breaking open of the surgical incision along the suture. Number of participants with dehiscence (reported as "yes") and number of participants showing no dehiscence (reported as "No").
Time Frame: At Day 10
Population: Analysis was performed on Full analysis set (FAS) that included all participants randomized that were allocated to one of the 2 treatment groups and had at least 1 post-treatment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 28 | 59
Participants
  No Dehiscence | 27 | 46
  Dehiscence | 1 | 13

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as any adverse event (AE) that occured during the on-treatment-period (i.e. after the start of the application of the Investigational Medical Device (IMD) (Day 0) until the end-of-treatment visit [Month 3]).This included any events related to the procedures, the IMD, or the comparator. An SAE was any untoward medical occurrence or effect that: led to death, or led to serious deterioration in the health of the participant, that either resulted in: life-threatening illness or injury, or a permanent impairment of a body structure or a body function, or in-patient or prolonged hospitalization, or medical or surgical intervention to prevent life-threatening illness or injury or permanent, or impairment to a body structure or a body function. Or, led to fetal distress, fetal death, or a congenital abnormality or birth defect.
Time Frame: From Baseline (Day 0) up to Month 3
Population: Analysis was performed on safety analysis set that included all participants where the application of MAR-CUTIS or Dermabond Advanced had started. Participants were analyzed under the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 29 | 60
Participants
  Any TEAE | 13 | 36
  Any serious TEAE | 4 | 13
  Any TEAE leading to withdrawal from trial | 0 | 2

3. Secondary Outcome: Number of Participants With Total Dehiscence of Target Wound at Month 1
Description: Wound dehiscence involved the breaking open of the surgical incision along the suture.
Time Frame: At Month 1
Population: Study was terminated early and data was not collected for this assessment.
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participant's Reporting Satisfaction With the Device Using Patient and Observer Scar Assessment Scale (POSAS)
Description: The POSAS was a questionnaire that was developed to assess scar quality. It consisted of 2 separate 6-item scales (Patient Scale and Observer Scale), both of which were scored on a 10-point rating scale. In addition, each scale has an overall "opinion" with 1 being no pain, no itching, or normal skin and 10 being worst scar imaginable with pain and itching, where lower scores indicated better outcome.
Time Frame: At Month 1 and Month 3
Population: Study was terminated early and data was not collected for this assessment.
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Wound Infections
Description: The wound infection incidence was assessed at the scheduled visits diagnosed according to the Centers for Disease Control and Prevention (CDC) criteria for surgical site infection. Wound infection was assessed and the following symptoms were evaluated if infection was present:
  * Presence of erythema
  * Presence of edema
  * Presence of pain at rest
  * Presence of elevated temperature
  Percentage of participants with wound infections around target wound are reported.
Time Frame: At Day 10, and Month 1
Population: Analysis was performed on FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 28 | 59
percentage of participants
  Day 10 | 0 | 3.4
  Month 1 | 0 | 3.4

6. Secondary Outcome: Investigator's Satisfaction With the Device Using Patient and Observer Scar Assessment Scale (POSAS)
Description: The POSAS was a questionnaire that was developed to assess scar quality. Investigator were asked to rate the severity of participant's scar compared to normal skin. The overall "opinion" ranged from 1= no pain, no itching, or normal skin to 10 = worst scar imaginable with pain and itching, where lower scores indicated better outcome.
Time Frame: At Month 1 and Month 3
Population: Study was terminated early and data was not collected for this assessment.
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Investigator's Satisfaction With the Device Using Modified Hollander Cosmesis Scale
Description: The investigator's satisfaction with the cosmetic outcome was assessed using the Modified Hollander Cosmesis Scale (mHCS). The mHCS consisted of 6 wound characteristics: Step-off borders, Contour irregularities, Target wound margin separation, Edge inversion, Excessive inflammation, Overall appearance. It was evaluated as "poor" or "good". Each of the characteristics was graded on a 0 (no/good) or 1 (yes/poor) point scale, where lower score indicated better outcome. Number of participants with different wound characteristics (poor and good) and participants with missing response are also reported.
Time Frame: At Day 10 and Month 1
Population: Analysis was performed on FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 28 | 59
Participants
  Day 10: Step-off borders: poor | 2 | 8
  Day 10: Step-off borders: good | 22 | 47
  Day 10: Step-off borders: missing | 4 | 4
  Day 10: Contour irregularities: poor | 2 | 9
  Day 10: Contour irregularities: good | 22 | 46
  Day 10: Contour irregularities: missing | 4 | 4
  Day 10: Wound margin separation: poor | 1 | 11
  Day 10: Wound margin separation: good | 23 | 44
  Day 10: Wound margin separation: missing | 4 | 4
  Day 10: Edge inversion: poor | 1 | 5
  Day 10: Edge inversion: good | 23 | 50
  Day 10: Edge inversion: missing | 4 | 4
  Day 10: Excessive inflammation: poor | 3 | 1
  Day 10: Excessive inflammation: good | 21 | 54
  Day 10: Excessive inflammation: missing | 4 | 4
  Day 10: Overall appearance: poor | 1 | 6
  Day 10: Overall appearance: good | 23 | 49
  Day 10: Overall appearance: Missing | 4 | 4
  Month 1: Step-off borders: poor | 0 | 3
  Month 1: Step-off borders: good | 25 | 50
  Month 1: Step-off borders: missing | 3 | 5
  Month 1: Contour irregularities: poor | 2 | 1
  Month 1: Contour irregularities: good | 23 | 52
  Month 1: Contour irregularities: missing | 3 | 5
  Month 1: Wound margin separation: poor | 1 | 5
  Month 1: Wound margin separation: good | 24 | 48
  Month 1: Wound margin separation: missing | 3 | 5
  Month 1: Edge inversion: poor | 1 | 1
  Month 1: Edge inversion: good | 24 | 52
  Month 1: Edge inversion: missing | 3 | 5
  Month 1: Excessive inflammation: poor | 1 | 2
  Month 1: Excessive inflammation: good | 24 | 51
  Month 1: Excessive inflammation: missing | 3 | 5
  Month 1: Overall appearance: poor | 0 | 3
  Month 1: Overall appearance: good | 25 | 50
  Month 1: Overall appearance: missing | 3 | 5

8. Secondary Outcome: Number of Participant Reporting Satisfaction With the Device Using a Product-Related Questionnaire
Description: The questionnaire consisted of 5 yes/no questions that evaluated the participant's experience with the adhesive, 1 question that rated the effect of the closed wound on several daily activities (i.e., showering, getting dressed), 1 question that evaluated satisfaction with the wound closure, and visual analog scales which rate pain and scarring.
Time Frame: At Day 10 and Month 1
Population: Study was terminated early and data was not collected for this assessment.
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Reporting Satisfaction With the Device Evaluated by Investigator Using a Product-Related Questionnaire
Description: The questionnaire consisted of 5 yes/no questions that assess the investigator's experience applying the adhesive (i.e., easy to use, fast, without complications), a visual analog scale that rates usability of the product from 1 (poor = very difficult to use) to 100 (excellent = very easy to use), and 1 question that evaluates satisfaction with the adhesive.
Time Frame: At Day 0 and Month 1
Population: Study was terminated early and data was not collected for this assessment.
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Investigator's Satisfaction With Ease of Use With the Device Using a Product-Related Questionnaire
Description: The questionnaire consisted of 8 yes/no questions and 1 opinion question that evaluated the investigator's experience with use of the adhesive (i.e., instructions easy to understand, preparation of the syringe being easy and fast, glue hardening time).
Time Frame: At Month 1
Population: Study was terminated early and data was not collected for this assessment.
Arm/Group | Dermabond Advanced | MAR-CUTIS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data was collected from Baseline until the end-of-treatment visit (Month 3).
Description: Reported AEs and deaths are TEAEs that was defined as any adverse event that occurred during the on-treatment-period (i.e. after the start of the application of the IMD (Baseline [Day 0]) until the end-of-treatment visit (Month 3). Analysis was performed on safety analysis set.
Arm/Group | Dermabond Advanced | MAR-CUTIS
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/60
Serious Adverse Events (participants affected / at risk) | 4/29 | 13/60
Other Adverse Events (participants affected / at risk) | 12/29 | 31/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dermabond Advanced (N=29) | MAR-CUTIS (N=60)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dermabond Advanced (N=29) | MAR-CUTIS (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 6 (8)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 6 (7)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (7)
Dehiscence (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 6 (6)
Swelling (General disorders) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 3 (3)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Drain site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 4 (4)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Cortisol decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Genital swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Itching scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to sponsor's discretion, as primary goal of the study could not be reached anymore at the time of termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any proposed presentation of the results of this trial before they are submitted for publication or public disclosure. Neither party (e.g., the sponsor, the coordinating investigator) has the right to prohibit publication or public disclosure unless it can be shown to affect possible patent rights.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT03688880/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT03688880/SAP_001.pdf